CLINICAL TRIAL: NCT03548259
Title: Effects of Platelet-rich Plasma in the Surgery of Carpal Tunnel Syndrome: A Randomized
Brief Title: Effects of Platelet-rich Plasma in the Surgery of Carpal Tunnel Syndrome: A Randomized Controlled Trial
Acronym: PRP-CTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-18
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Platelet-rich plasma; Surgery
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (Parallel Assignment)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Platelet-rich plasma
  Interventions: Procedure: Platelet-rich plasma; Procedure: Platelet-poor plasma
- Platelet-poor plasma (Placebo Comparator): Platelet-poor plasma
  Interventions: Procedure: Platelet-rich plasma; Procedure: Platelet-poor plasma

INTERVENTIONS:
Procedure: Platelet-rich plasma — Platelet-rich plasma injection
Procedure: Platelet-poor plasma — Platelet-poor plasma injection

SUMMARY:
The Platelet-rich plasma (PRP) has been proved to be efficient in the non-surgical treatment of carpal tunnel syndrome (CTS). Here we propose to assess the effectiveness of PRP as co-adjuvant in surgical treatment of CTS by open carpal tunnel release.

Design: Randomized Controlled Trial. Setting: Local Hospital.

DETAILED DESCRIPTION:
Carpal tunnel syndrome (CTS) is a common disorder with an estimated annual incidence of 125-542 in adults, and an estimated prevalence of 1 to 5 percent in the general population. CTS is the most frequent compressive focal mononeuropathy and causes pain, paresthesia and weakness of the median nerve distribution in patients.

The treatment of the CTS includes both, conservative and surgical treatment depending on the severity of the symptoms.

Platelet-rich plasma (PRP) has been proved to be efficient in the non-surgical treatment of CTS, however its potential used as co-adjuvant in surgical treatment has not been assessed.

We propose a randomized clinical trial in patients in which the surgical treatment is indicated. Participants in the intervention group receive a PRP injection, and in the control group a platelet-poor plasma injection after open carpal tunnel release. The evaluation is performed pretreatment as well as on the 6st week after treatment. Outcome measures include: hand grip strength (primary outcome), pain, sympton severity and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Carpal Tunnel Syndrome (CTS)
* Conservative treatment failure

Exclusion Criteria:

* Previous CTS surgery on the same side
* Wrist fracture/trauma in history
* Polyneuropathy
* Diabetes mellitus
* Cervical neuropathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 6 weeks
  Hand grip strength measured with dynamometer

SECONDARY OUTCOMES:
Pain | 6 weeks
  Pain measured with the Wong-Baker Faces Pain Rating Scale. The scale shows a series of faces ranging from a happy face at 0 which represents "no hurt" to a crying face at 10 which represents "hurts worst".
Sympton severity | 6 weeks
  Sympton severity measured with the sympton severity scale of the Boston Carpal Tunnel Syndrome Questionnaire. The Symptom Severity Scale (SSS) contains 11 questions and uses a five-point rating scale that generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.
Functional status | 6 weeks
  Functional status measured with the sympton severity scale of the Boston Carpal Tunnel Syndrome Questionnaire.The Functional Status Scale (FSS) contains 8 items and uses a five-point rating scale that generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.
Wound healing | 6 weeks
  Wound healing measured with the Southampton Wound Assessment Scale. Wounds are scored as 0, I, II, III, IV and V, with a higher score indicating worst healing.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Pérez, PhD, Study Chair — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided